CLINICAL TRIAL: NCT03609957
Title: Effect of Exercise on Pain Responses in Non-Hispanic Blacks and Whites
Brief Title: Exercise and Pain in Non-Hispanic Blacks and Whites
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Did not have time to complete this study
Sponsor: Georgia State University (Other)
Responsible Party: Principal Investigator, Brett Wong, Principal Investigator, Georgia State University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: R01HL141205 (NIH)
Record Dates: First submitted 2018-07-11; First posted 2018-08-01 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Pain, Acute; Pain, Neuropathic; Analgesia; Aerobic Exercise; Exercise Training
MeSH Terms: conditions — Acute Pain; Neuralgia; Agnosia | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic Exercise Training (Experimental): Moderate intensity (75% heart rate reserve) cycling exercise for 32 minutes, 3 days per week for 5 weeks
  Interventions: Other: Aerobic Exercise Training
- Interval Training (Experimental): High intensity (95% heart rate reserve) cycling exercise for 20 minutes, 3 days per week for 5 weeks
  Interventions: Other: Interval Training
- Control (No Intervention): Control (no exercise intervention) group

INTERVENTIONS:
Other: Aerobic Exercise Training — Traditional, continuous aerobic exercise (cycling) at a moderate intensity
  Arms: Aerobic Exercise Training
Other: Interval Training — High-intensity interval exercise consisting of short bursts of exercise interspersed with rest periods
  Arms: Interval Training

SUMMARY:
Non-Hispanic Blacks tend to report higher levels of pain, experience pain more frequently, and be under-treated for pain compared to non-Hispanic Whites. Acute (single session) exercise is known to be effective at reducing pain but it is unknown what effect chronic exercise training has on pain responses. The broad goal of this study is to determine whether regular exercise training is more effective at reducing pain responses in non-Hispanic Blacks compared to non-Hispanic Whites. The investigators are interested in comparing regular aerobic exercise training versus high-intensity interval training.

DETAILED DESCRIPTION:
Racial discrepancy in the experience of pain is well documented within the literature. Non-Hispanic Blacks (NHB) report greater amounts and severity of clinical pain compared to non-Hispanic Whites (NHW) in a variety of clinical conditions. NHB also experience greater pain-related symptoms and disability, regardless of descriptive factors such as age, gender, and socioeconomic status or clinical factors such as comorbidities and duration of disease. Further, NHB tend to be medically undertreated for pain, regardless of nearly identical reporting of pain level and severity compared with NHW. Not only is adequate pain treatment infrequent, but many pain treatments are less effective in NHB than in NHW, commonly resulting in less reduction of pain severity in this population.

In comparison to NHW, NHB report greater sensitivity to several types of pain, including heat pain, cold pressor pain, ischemic pain, and electrical stimulation. NHB show increased temporal summation, implying central nervous system hypersensitivity and hyperexcitability to noxious (painful) stimuli. Specifically, regarding experimental heat pain, NHB differ minimally in pain threshold or ratings of pain intensity compared to NHW, but perceive greater unpleasantness of pain and show a lower pain tolerance. The physiological mechanisms underlying this racial discrepancy remain unknown.

Experimental pain assessment is valuable in understanding the experience of pain between individuals. Pain is an individual experience and differs from one to another. However, differences in experimental pain perceived may estimate the clinical pain one would experience. Studies show that greater experimental pain sensitivity is associated with greater experience of day-to-day pain in healthy adults and can predict higher levels of clinical pain in adult patients.

While affective (subjective) pain perception has been the focus of the majority of pain assessment studies, in 2008 Campbell et al. investigated the nociceptive flexion reflex (NFR), an involuntary and objective component of the pain response. The NFR is a spinal-mediated reflex that follows activation of nociceptive A-delta afferents by noxious stimuli. This study shows the NFR threshold in NHB is decreased compared to NHW, implying a physiological difference between these racial groups that may contribute to the discrepancy in pain perception. Skin blood flow via vasodilation, another physiological measure, has been shown to increase in response to noxious thermal stimuli in order to distribute heat away from a singular point in the cutaneous environment and prevent damage. Assessing changes in skin blood flow in response to noxious thermal stimuli may further elucidate physiological differences between races that affect pain perception.

It is important to investigate more effective prevention or treatment methods for pain in NHB. Exercise-induced hypoalgesia (EIH) is characterized by decreased pain sensation following physical exercise. Specifically, EIH leads to decreased sensitivity to noxious (painful) stimuli, increased pain thresholds, increased pain tolerance, and decreased pain ratings. EIH has been shown to occur following several types of exercise, such as acute bouts of submaximal, continuous aerobic exercise and acute bouts of isometric hand-grip exercise. Lending to the knowledge of racial discrepancy in pain perception, a study by Umeda et al. in 2016 showed NHB had a smaller magnitude of EIH compared to NHW following isometric hand-grip exercise, but racial differences in EIH remain incompletely understood.

It is suggested that hypoalgesia following exercise may be due to an overlapping of pain perception and cardiovascular mechanisms. For example, pain regulation and blood pressure control are associated with the same brain stem nuclei. Further, hypertensive individuals have shown reduced sensitivity to noxious (painful) stimuli compared to normotensives, and acute pharmacological elevations in blood pressure have been shown to alter pain perception. Therefore, it is important to investigate alterations in pain perception following both acute (which should elicit elevations in blood pressure) and chronic (which should elicit overall declines in blood pressure) exercise.

Several studies have investigated the effects of submaximal exercise on various types of pain and it is typical to see moderate-intensity continuous (MIC) exercise incorporated into pain management programs (generally 30 minutes of 70% VO2max exercise). However, two studies in particular display data indicating that as workload increases, pain thresholds increase in a stepwise manner. Other studies show EIH occurs more consistently following exercise at higher intensities (> 70% VO2max), indicating that high intensity interval training (HIIT) may produce more beneficial results in affective and/or objective responses to pain than MIC exercise. Several studies have looked at affective pain perception following acute submaximal bouts of aerobic and isometric exercise. Those that have investigated acute HIIT have only examined affective responses. The investigators do not know of any studies that have looked at the acute and chronic effect of MIC exercise and HIIT on affective and objective pain perception in NHB and NH There are three main purposes of this study, and they are as follows: 1) to assess objective and subjective responses to pain in NHB and NHW, 2) to assess the use of acute versus chronic exercise in pain management for NHW and NHB, and 3) to assess the use of MIC exercise versus HITT in pain management for NHW and NHB. The investigators hypothesize that 1) NHB will show decreased skin blood flow response to noxious stimuli compared to NHW prior to exercise training, 2) NHB will report greater pain ratings than NHW prior to exercise training, and 3) chronic HIIT will mitigate the differences in skin blood flow and pain ratings between NHB and NHW.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Normotensive
* Identify as non-Hispanic Black or non-Hispanic White
* Healthy enough to participate in regular exercise
* Not taking any medications other than birth control

Exclusion Criteria:

* Heart disease (high blood pressure, previous stroke or heart attack)
* Type 1 or 2 diabetes
* History of cancer treated with chemotherapy
* History of nerve damage
* History of chronic pain
* Current smoker/tobacco user or quit less than 1 year ago
* Skin disorders (psoriasis, etc.)
* Pregnant
* Taking any medications other than birth control

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change in skin blood flow response to local heating | Baseline (prior to intervention or control) and at the conclusion of the 5-week intervention or control. The post-intervention assessment will be performed no later than 3-5 days after completion of the 5-week intervention or control.
  Vasodilation in response to painful and non-painful heating of the skin

CONTACTS AND LOCATIONS:
Overall Officials: Brett J Wong, Ph.D., Principal Investigator — Georgia State University
Locations (1):
- Georgia State University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
The current approved IRB and informed consent state that we will not share participants' data except with applicable oversight bodies (IRB, FDA, OHRP, etc.).

REFERENCES:
- [Background] Green CR, Anderson KO, Baker TA, Campbell LC, Decker S, Fillingim RB, Kalauokalani DA, Lasch KE, Myers C, Tait RC, Todd KH, Vallerand AH. The unequal burden of pain: confronting racial and ethnic disparities in pain. Pain Med. 2003 Sep;4(3):277-94. doi: 10.1046/j.1526-4637.2003.03034.x. PMID 12974827
- [Background] Klonoff EA. Disparities in the provision of medical care: an outcome in search of an explanation. J Behav Med. 2009 Feb;32(1):48-63. doi: 10.1007/s10865-008-9192-1. Epub 2009 Jan 6. PMID 19127421
- [Background] Riley JL 3rd, Wade JB, Myers CD, Sheffield D, Papas RK, Price DD. Racial/ethnic differences in the experience of chronic pain. Pain. 2002 Dec;100(3):291-298. doi: 10.1016/S0304-3959(02)00306-8. PMID 12468000
- [Background] Edwards RR, Doleys DM, Fillingim RB, Lowery D. Ethnic differences in pain tolerance: clinical implications in a chronic pain population. Psychosom Med. 2001 Mar-Apr;63(2):316-23. doi: 10.1097/00006842-200103000-00018. PMID 11292281
- [Background] Green CR, Baker TA, Sato Y, Washington TL, Smith EM. Race and chronic pain: A comparative study of young black and white Americans presenting for management. J Pain. 2003 May;4(4):176-83. doi: 10.1016/s1526-5900(02)65013-8. PMID 14622701
- [Background] Bruce B, Fries JF, Murtagh KN. Health status disparities in ethnic minority patients with rheumatoid arthritis: a cross-sectional study. J Rheumatol. 2007 Jul;34(7):1475-9. Epub 2007 Jun 1. PMID 17552045
- [Background] Cano A, Mayo A, Ventimiglia M. Coping, pain severity, interference, and disability: the potential mediating and moderating roles of race and education. J Pain. 2006 Jul;7(7):459-68. doi: 10.1016/j.jpain.2006.01.445. PMID 16814685
- [Background] Golightly YM, Dominick KL. Racial variations in self-reported osteoarthritis symptom severity among veterans. Aging Clin Exp Res. 2005 Aug;17(4):264-9. doi: 10.1007/BF03324608. PMID 16285190
- [Background] Vallerand AH, Hasenau S, Templin T, Collins-Bohler D. Disparities between black and white patients with cancer pain: the effect of perception of control over pain. Pain Med. 2005 May-Jun;6(3):242-50. doi: 10.1111/j.1526-4637.2005.05038.x. PMID 15972088
- [Background] Mechlin B, Heymen S, Edwards CL, Girdler SS. Ethnic differences in cardiovascular-somatosensory interactions and in the central processing of noxious stimuli. Psychophysiology. 2011 Jun;48(6):762-73. doi: 10.1111/j.1469-8986.2010.01140.x. Epub 2010 Oct 29. PMID 21039586
- [Background] Anderson KO, Mendoza TR, Valero V, Richman SP, Russell C, Hurley J, DeLeon C, Washington P, Palos G, Payne R, Cleeland CS. Minority cancer patients and their providers: pain management attitudes and practice. Cancer. 2000 Apr 15;88(8):1929-38. PMID 10760771
- [Background] Merry B, Campbell CM, Buenaver LF, McGuire L, Haythornthwaite JA, Doleys DM, Edwards RR. Ethnic Group Differences in the Outcomes of Multidisciplinary Pain Treatment. J Musculoskelet Pain. 2011 Jan;19(1):24-30. doi: 10.3109/10582452.2010.538821. PMID 21731407
- [Background] Siedlecki SL. Racial variation in response to music in a sample of African-American and Caucasian chronic pain patients. Pain Manag Nurs. 2009 Mar;10(1):14-21. doi: 10.1016/j.pmn.2008.08.003. PMID 19264279
- [Background] Campbell CM, Edwards RR, Fillingim RB. Ethnic differences in responses to multiple experimental pain stimuli. Pain. 2005 Jan;113(1-2):20-6. doi: 10.1016/j.pain.2004.08.013. PMID 15621360
- [Background] Chapman WP, Jones CM. VARIATIONS IN CUTANEOUS AND VISCERAL PAIN SENSITIVITY IN NORMAL SUBJECTS. J Clin Invest. 1944 Jan;23(1):81-91. doi: 10.1172/JCI101475. No abstract available. PMID 16695086
- [Background] Sheffield D, Biles PL, Orom H, Maixner W, Sheps DS. Race and sex differences in cutaneous pain perception. Psychosom Med. 2000 Jul-Aug;62(4):517-23. doi: 10.1097/00006842-200007000-00010. PMID 10949097
- [Background] Edwards RR, Fillingim RB. Ethnic differences in thermal pain responses. Psychosom Med. 1999 May-Jun;61(3):346-54. doi: 10.1097/00006842-199905000-00014. PMID 10367615
- [Background] Walsh NE, Schoenfeld L, Ramamurthy S, Hoffman J. Normative model for cold pressor test. Am J Phys Med Rehabil. 1989 Feb;68(1):6-11. doi: 10.1097/00002060-198902000-00003. PMID 2917058
- [Background] Campbell CM, France CR, Robinson ME, Logan HL, Geffken GR, Fillingim RB. Ethnic differences in the nociceptive flexion reflex (NFR). Pain. 2008 Jan;134(1-2):91-6. doi: 10.1016/j.pain.2007.03.035. Epub 2007 May 4. PMID 17482362
- [Background] Campbell CM, Edwards RR. Ethnic differences in pain and pain management. Pain Manag. 2012 May;2(3):219-230. doi: 10.2217/pmt.12.7. PMID 23687518
- [Background] Clauw DJ, Williams D, Lauerman W, Dahlman M, Aslami A, Nachemson AL, Kobrine AI, Wiesel SW. Pain sensitivity as a correlate of clinical status in individuals with chronic low back pain. Spine (Phila Pa 1976). 1999 Oct 1;24(19):2035-41. doi: 10.1097/00007632-199910010-00013. PMID 10528381
- [Background] Fillingim RB, Maixner W, Kincaid S, Sigurdsson A, Harris MB. Pain sensitivity in patients with temporomandibular disorders: relationship to clinical and psychosocial factors. Clin J Pain. 1996 Dec;12(4):260-9. doi: 10.1097/00002508-199612000-00005. PMID 8969871
- [Background] Langemark M, Jensen K, Jensen TS, Olesen J. Pressure pain thresholds and thermal nociceptive thresholds in chronic tension-type headache. Pain. 1989 Aug;38(2):203-10. doi: 10.1016/0304-3959(89)90239-x. PMID 2780074
- [Background] Edwards RR, Fillingim RB. Age-associated differences in responses to noxious stimuli. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M180-5. doi: 10.1093/gerona/56.3.m180. PMID 11253160
- [Background] Fillingim RB, Edwards RR, Powell T. The relationship of sex and clinical pain to experimental pain responses. Pain. 1999 Dec;83(3):419-425. doi: 10.1016/S0304-3959(99)00128-1. PMID 10568849
- [Background] Kellogg DL Jr, Liu Y, Kosiba IF, O'Donnell D. Role of nitric oxide in the vascular effects of local warming of the skin in humans. J Appl Physiol (1985). 1999 Apr;86(4):1185-90. doi: 10.1152/jappl.1999.86.4.1185. PMID 10194201
- [Background] Koltyn KF, Umeda M. Exercise, hypoalgesia and blood pressure. Sports Med. 2006;36(3):207-14. doi: 10.2165/00007256-200636030-00003. PMID 16526833
- [Background] Pertovaara A, Huopaniemi T, Virtanen A, Johansson G. The influence of exercise on dental pain thresholds and the release of stress hormones. Physiol Behav. 1984 Dec;33(6):923-6. doi: 10.1016/0031-9384(84)90230-0. PMID 6100393
- [Background] Janal MN, Colt EWD, Clark CW, Glusman M. Pain sensitivity, mood and plasma endocrine levels in man following long-distance running: effects of naloxone. Pain. 1984 May;19(1):13-25. doi: 10.1016/0304-3959(84)90061-7. PMID 6330643
- [Background] Kemppainen P. Modification of human dental pain thresholds by conditioning stimulation. Proc Finn Dent Soc. 1985;81 3-4:1-67. No abstract available. PMID 3832067
- [Background] Koltyn KF, Garvin AW, Gardiner RL, Nelson TF. Perception of pain following aerobic exercise. Med Sci Sports Exerc. 1996 Nov;28(11):1418-21. doi: 10.1097/00005768-199611000-00011. PMID 8933493
- [Background] Gurevich M, Kohn PM, Davis C. Exercise-induced analgesia and the role of reactivity in pain sensitivity. J Sports Sci. 1994 Dec;12(6):549-59. doi: 10.1080/02640419408732205. PMID 7853451
- [Background] Bartholomew JB, Lewis BP, Linder DE, Cook DB. Post-exercise analgesia: replication and extension. J Sports Sci. 1996 Aug;14(4):329-34. doi: 10.1080/02640419608727718. PMID 8887212
- [Background] Kemppainen P, Hamalainen O, Kononen M. Different effects of physical exercise on cold pain sensitivity in fighter pilots with and without the history of acute in-flight neck pain attacks. Med Sci Sports Exerc. 1998 Apr;30(4):577-82. doi: 10.1097/00005768-199804000-00016. PMID 9565940
- [Background] Vierck CJ Jr, Staud R, Price DD, Cannon RL, Mauderli AP, Martin AD. The effect of maximal exercise on temporal summation of second pain (windup) in patients with fibromyalgia syndrome. J Pain. 2001 Dec;2(6):334-44. doi: 10.1054/jpai.2001.25533. PMID 14622813
- [Background] Koltyn KF. Analgesia following exercise: a review. Sports Med. 2000 Feb;29(2):85-98. doi: 10.2165/00007256-200029020-00002. PMID 10701712
- [Background] Umeda M, Kempka LE, Greenlee BT, Weatherby AC. A smaller magnitude of exercise-induced hypoalgesia in African Americans compared to non-Hispanic Whites: A potential influence of physical activity. Biol Psychol. 2016 Jan;113:46-51. doi: 10.1016/j.biopsycho.2015.11.006. Epub 2015 Nov 28. PMID 26607443
- [Background] Ghione S. Hypertension-associated hypalgesia. Evidence in experimental animals and humans, pathophysiological mechanisms, and potential clinical consequences. Hypertension. 1996 Sep;28(3):494-504. doi: 10.1161/01.hyp.28.3.494. PMID 8794839
- [Background] Lovick TA. Integrated activity of cardiovascular and pain regulatory systems: role in adaptive behavioural responses. Prog Neurobiol. 1993 May;40(5):631-44. doi: 10.1016/0301-0082(93)90036-r. No abstract available. PMID 8484005
- [Background] Zamir N, Maixner W. The relationship between cardiovascular and pain regulatory systems. Ann N Y Acad Sci. 1986;467:371-84. doi: 10.1111/j.1749-6632.1986.tb14641.x. PMID 3524385
- [Background] France CR. Decreased pain perception and risk for hypertension: considering a common physiological mechanism. Psychophysiology. 1999 Nov;36(6):683-92. PMID 10554582
- [Background] Koltyn KF. Exercise-induced hypoalgesia and intensity of exercise. Sports Med. 2002;32(8):477-87. doi: 10.2165/00007256-200232080-00001. PMID 12076175
- [Background] Kemppainen P, Pertovaara A, Huopaniemi T, Johansson G, Karonen SL. Modification of dental pain and cutaneous thermal sensitivity by physical exercise in man. Brain Res. 1985 Dec 23;360(1-2):33-40. doi: 10.1016/0006-8993(85)91217-x. PMID 3000534
- [Background] Kodesh E, Weissman-Fogel I. Exercise-induced hypoalgesia - interval versus continuous mode. Appl Physiol Nutr Metab. 2014 Jul;39(7):829-34. doi: 10.1139/apnm-2013-0481. Epub 2014 Feb 12. PMID 24773287